CLINICAL TRIAL: NCT05970692
Title: Cross-Cultural Adaptation and Psychometric Validation of the Turkish Version of Atroshi-Lyrén 6-item Symptoms Scale
Status: Recruiting | Type: Observational
Sponsor: Ilke KARA (Other)
Collaborators: Bitlis Eren University (Other)
Responsible Party: Sponsor-Investigator, Ilke KARA, Co-Principal Investigator, Dokuz Eylul University
Organization: Dokuz Eylul University (Other)
Other Study IDs: BEU-KTS-01
Record Dates: First submitted 2023-07-24; First posted 2023-08-01 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Carpal Tunnel Syndrome
Keywords: Carpal Tunnel Syndrome; Pain
MeSH Terms: conditions — Carpal Tunnel Syndrome; Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Controls: Healthy individuals aged between 18-65 years old
- CTS Group: CTS patients aged between 18-65 years old

SUMMARY:
This study aims to develop Turkish version of the Atroshi-Lyrén 6-item symptoms scale (A-L scale) and to perform validity and reliability evaluations.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18-65 years old,
* Had symptoms of numbness, tingling, weakness and pain in the hands for at least 1 month,
* Assessed through provocation tests and physical examination to match the median nerve distribution.

Exclusion Criteria:

* Not willing to participate in the study,
* Clinical or electrophysiological signs of proximal nerve compression,
* Diabetes or other metabolic disease,
* Rheumatoid arthritis or other general inflammatory diseases.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: CTS patients aged between 18-65 years old
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-09-26 (Actual); Primary Completion 2024-08-13 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Atroshi-Lyrén 6-item symptoms scale | 1 week
  The A-L scale consists of 6 items that inquire about severity and frequency of night and daytime numbness and tingling and pain. For each patient the item responses are scored from 1 (best) to5 (worst) and then averaged for the 6 items to yield a total score (only 1 missing item response is allowed)

CONTACTS AND LOCATIONS:
Locations (1):
- Bitlis Eren University, Bitlis, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided